CLINICAL TRIAL: NCT02769169
Title: Double-dose Ranibizumab for Polypoidal Choroidal Vasculopathy: A Prospective Randomized Multicenter Study
Brief Title: Double-dose Ranibizumab for Polypoidal Choroidal Vasculopathy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: study protocol changed
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Lu, MD, PhD，Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DREAM STUDY
Record Dates: First submitted 2016-05-01; First posted 2016-05-11 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Ranibizumab, regression of the polyps
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- double-dose (Experimental): double-dose
  Lucentis® (Raibizumab), 1mg, 3+prn
  Interventions: Drug: Lucentis® (Raibizumab) double-dose
- regular-dose (Active Comparator): regular-dose
  Lucentis® (Raibizumab), 0.5mg, 3+prn
  Interventions: Drug: Lucentis® (Raibizumab) regular-dose

INTERVENTIONS:
Drug: Lucentis® (Raibizumab) double-dose — Give patients 1 injection per month at the beginning 3 months. Give patients additional injection as needed. One injection contains 1mg of Lucentis® (Raibizumab). Intervention 'double-dose: Ranibizumab 1mg, 3 injection plus prn' has not been included in any Arm/Group Descriptions.
  Arms: double-dose
Drug: Lucentis® (Raibizumab) regular-dose — Give patients 1 injection per month at the beginning 3 months. Give patients additional injection as needed. One injection contains 0.5mg of Lucentis® (Raibizumab). regular-dose: Ranibizumab 0.5mg, 3 injection plus prn
  Arms: regular-dose

SUMMARY:
The purpose of this study is to determine whether double-dose Ranibizumab are effective to regress the polyps and benefit to the visual outcome in the polypoidal choroidal vasculopathy (PCV).

DETAILED DESCRIPTION:
Recently, it's reported that intravitreal high dose Lucentis®（Ranibizumab） could benefit to both regression of the polyps and the relief of macular edema in PCV patients. Since it was a single arm prospective study with a relatively small sample size, randomized clinical trials were needed to confirm the efficacy of high dose Ranibizumab in PCV treatment. In this study, the investigator will compare the efficacy of double-dose (1mg, 3+prn) Raibizumab with regular dose (0.5mg, 3+prn) for PCV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years and ≤80;
* Active PCV confirmed by ICGA+FFA (Indocyanine green angiography + fundus fluorescein angiography);
* At least one distinguishable polyp was shown in ICGA;
* BCVA between 24 to 73 letters with ETDRS chart (Early Treatment of Diabetic Retinopathty Study);
* The greatest linear dimension of the lesion <5400μm.

Exclusion Criteria:

* Previously received treatment of laser retina photocoagulation, transpupillary thermotherapy, pneumatic displacement of subretinal blood or any investigational treatment;
* Previous photodynamic therapy or anti-Vegf treatment within 6 months in study eye
* Previously received treatment of photodynamic treatment within 1 month, or any anti-vascular endothelial growth factor (VEGF) intraocular injection in 3 months in the fellow eye;
* Combine of current vitreous hemorrhage or extensive subretinal hemorrhage (lesion area >30mm2);
* A history of angioid streaks, presumed ocular histoplasmosis syndrome or pathologic myopia;
* Experienced retinal pigmental epithelium (RPE) tear, retinal detachment, macular hole or uncontrolled glaucoma;
* Undergone intraocular surgery (except uncomplicated cataract extraction with intraocular lens implantation);
* Cataract extraction with intraocular lens implantation within 60 days;
* Combine of cataract that could require medical or surgical intervention during 12 months;
* Combine of diabetes mellitus and have poor glucose control (Haemoglobin A1c (HbA1c) >8%);
* Combine of hypertension and have poor blood pressure control (blood pressure ≥140/95 mmHg after regular antihypertensive drugs treatment);
* History of myocardial infarction or cerebral infarction in last 6 months;
* During gestation period or lactation period;
* Combine of confirmed systemic autoimmune disease or any uncontrollable clinical conditions (e.g. HIV, malignant tumor, active hepatitis, severe systemic disease, diseases need immediately surgical treatment).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants who have at least 1 polyp resolution | 6 months
  Number of participants who have at least 1 polyp resolution, assessed by Indocyanine angiography (ICGA) between baseline and Month 6

SECONDARY OUTCOMES:
change of best corrected visual acuity(BCVA) | Baseline to 6 months
  Mean change in BCVA, from baseline to the end of 6 month. As assessed by changes of number of letters with the ETDRS (Early Treatment of Diabetic Retinopathy Study) chart
change of central foveal thickness | Baseline to 6 months
  Mean change of central foveal thickness, from baseline to the end of 6 month. As assessed by optical coherence tomography scanning
Injection frequency | Baseline to 6 months
  Average injection number(from baseline to the end of 6 month), assessed by the number of intravitreal injection from baseline to month 6
Safety analysis: number of adverse event | 6 months
  Serious ocular adverse events in the study eye, including reduced VA, retinal hemorrhage, endophthalmitis, corneal edema, iridocyclitis, macular degeneration, retinal artery occlusion, retinal tear, retinal vein occlusion and vitreous floaters. Antiplatelet Trialists' Collaboration (APTC) arterial thromboembolic events (ATEs): including deaths (vascular or unknown cause), nonfatal myocardial infarction and hemorrhagic or ischemic nonfatal cerebrovascular accident. Serious adverse event of special interest, including ATE, bleeding/hemorrhage in central nervous system (CNS) or non-CNS, congestive heart failure, fistulae, gastrointestinal perforation, hypertension, venous thrombotic events and wound healing complications.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, MD, phD, Principal Investigator — Zhongshan Ophthalmic Center Guangzhou, Guangdong China
Locations (4):
- China (4):
  - Zhongshan Ophthalmic Center Guangzhou, Guangzhou, Guangdong
  - Retina surgery department, Shenzhen Eye Hospital of Second Clinical Medical College of Jinan University, Shenzhen, Guangdong
  - The First People's Hospital of Xuzhou, Xuzhou, Jiangsu
  - Dept. of Ophthalmology，Minhang hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Busbee BG, Ho AC, Brown DM, Heier JS, Suner IJ, Li Z, Rubio RG, Lai P; HARBOR Study Group. Twelve-month efficacy and safety of 0.5 mg or 2.0 mg ranibizumab in patients with subfoveal neovascular age-related macular degeneration. Ophthalmology. 2013 May;120(5):1046-56. doi: 10.1016/j.ophtha.2012.10.014. Epub 2013 Jan 23. PMID 23352196
- [Result] Koh A, Lee WK, Chen LJ, Chen SJ, Hashad Y, Kim H, Lai TY, Pilz S, Ruamviboonsuk P, Tokaji E, Weisberger A, Lim TH. EVEREST study: efficacy and safety of verteporfin photodynamic therapy in combination with ranibizumab or alone versus ranibizumab monotherapy in patients with symptomatic macular polypoidal choroidal vasculopathy. Retina. 2012 Sep;32(8):1453-64. doi: 10.1097/IAE.0b013e31824f91e8. PMID 22426346
- [Result] Kokame GT. Prospective evaluation of subretinal vessel location in polypoidal choroidal vasculopathy (PCV) and response of hemorrhagic and exudative PCV to high-dose antiangiogenic therapy (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2014 Jul;112:74-93. PMID 25646029
- [Result] Kokame GT, Yeung L, Lai JC. Continuous anti-VEGF treatment with ranibizumab for polypoidal choroidal vasculopathy: 6-month results. Br J Ophthalmol. 2010 Mar;94(3):297-301. doi: 10.1136/bjo.2008.150029. Epub 2009 Sep 1. PMID 19726427
- [Result] Obata R, Yanagi Y, Kami J, Takahashi H, Inoue Y, Tamaki Y. Polypoidal choroidal vasculopathy and retinochoroidal anastomosis in Japanese patients eligible for photodynamic therapy for exudative age-related macular degeneration. Jpn J Ophthalmol. 2006 Jul-Aug;50(4):354-360. doi: 10.1007/s10384-005-0337-2. PMID 16897221
- [Result] Sho K, Takahashi K, Yamada H, Wada M, Nagai Y, Otsuji T, Nishikawa M, Mitsuma Y, Yamazaki Y, Matsumura M, Uyama M. Polypoidal choroidal vasculopathy: incidence, demographic features, and clinical characteristics. Arch Ophthalmol. 2003 Oct;121(10):1392-6. doi: 10.1001/archopht.121.10.1392. PMID 14557174